CLINICAL TRIAL: NCT05030428
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Trial, Assessing the Impact of Inclisiran on Major Adverse Cardiovascular Events in Participants With Established Cardiovascular Disease (VICTORION-2 PREVENT)
Brief Title: Study of Inclisiran to Prevent Cardiovascular (CV) Events in Participants With Established Cardiovascular Disease
Acronym: VICTORION-2P
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKJX839B12302
Record Dates: First submitted 2021-08-17; First posted 2021-09-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Atherosclerotic cardiovascular disease; Hypercholesterolemia; Dyslipidemia; high cholesterol; Hyperlipidemia; Inclisiran; siRNA; KJX839
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Dyslipidemias; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, parallel group, placebo-controlled, multi-center, event-driven study
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran sodium (Experimental): Subcutaneous injection
  Interventions: Drug: Inclisiran sodium 300 mg
- Placebo (Placebo Comparator): Subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclisiran sodium 300 mg — Subcutaneously injected on Day 1, Month 3 (Day 90) and every 6 months thereafter until EOS visit
  Arms: Inclisiran sodium
Drug: Placebo — Subcutaneously injected on Day 1, Month 3 (Day 90) and every 6 months thereafter until EOS visit
  Arms: Placebo

SUMMARY:
Study CKJX839B12302 is a pivotal Phase III trial to evaluate the benefits of inclisiran on major adverse cardiovascular (MACE) events in participants with established cardiovascular disease (CVD).

DETAILED DESCRIPTION:
Purpose of this study is to test the hypothesis that treatment with inclisiran sodium 300 mg s.c. administered on Day 1, Month 3 (Day 90), and every 6 months thereafter taken in addition to well-tolerated high-intensity statin therapy in participants with established ASCVD will significantly reduce the risk of 3-Point-Major Adverse Cardiovascular Events (3P-MACE) defined as a composite of CV death, non-fatal myocardial infarction (MI) and non-fatal ischemic stroke. This will be compared to placebo in adjunct to well-tolerated high-intensity statin therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Fasting LDL-C ≥ 70 mg/dL at randomization visit
2. Stable (greater than or equal to 4 weeks) and well-tolerated lipid-lowering regimen (including e.g. with or without Ezetimibe) that must include a high-intensity statin therapy with either atorvastatin greater than or equal to 40 mg QD or rosuvastatin greater than or equal to 20 mg QD
3. Established CV disease defined as ANY of the following three conditions

   1. Spontaneous Myocardial infarction ≥ 4 weeks from screening visit
   2. History of ischemic stroke occurred ≥ 4 weeks prior to the Screening visit
   3. Symptomatic peripheral arterial disease (PAD) evidenced by either intermittent claudication with ankle brachial index (ABI) < 0.85, prior peripheral arterial revascularization procedure, or, amputation due to atherosclerotic disease.

Exclusion Criteria:

1. Acute coronary syndrome, stroke, peripheral arterial revascularization procedure or amputation due to atherosclerotic disease < 4 weeks before screening visit
2. Treatment with PCSK9 inhibitors (e.g. evolocumab, alirocumab) within 90 days or planned use post first study visit
3. Planned or expected cardiac, cerebrovascular or peripheral artery surgery or re-vascularization within the 6 months after the first study visit
4. Heart failure NYHA class III or IV
5. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver
6. Previous exposure to inclisiran or any other non-mAb PCSK9-targeted therapy, either as an investigational or marketed drug within 2 years
7. Severe concomitant non-CV disease that is expected to reduce life expectancy to less than 5 years
8. History of malignancy that required surgery radiation therapy and/or systemic therapy during the 3 years prior to the first study visit
9. Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17004 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2027-10-13 (Estimated); Study Completion 2027-10-13 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of 3P-MACE (3-Point Major Adverse Cardiovascular Events) | From randomization to total follow-up time (up to 72 months)
  3P-MACE is a confirmed composite endpoint which includes cardiovascular death, non-fatal myocardial infarction and non-fatal ischemic stroke.

SECONDARY OUTCOMES:
Time to Occurrence of Cardiovascular (CV) Death | From randomization to total follow-up time (up to 72 months)
  CV death is defined as death due to cardiovascular events
Time to First Occurrence of 4P-MACE (4-Point Major Adverse Cardiovascular Events) | From randomization to total follow-up time (up to 72 months)
  A composite 4P- MACE is defined as CV death, non-fatal MI, non-fatal ischemic stroke and urgent coronary revascularization.
Time to first occurrence of Major Limb Adverse Events (MALE) | From randomization to total follow-up time (up to 72 months)
  Major Limb Adverse Events including acute lower limb ischemia, lower limb amputation due to ischemia, or urgent lower limb revascularization for ischemia
Time to occurrence of all-cause death | From randomization to total follow-up time (up to 72 months)
  All-Cause death is defined as: all deaths from randomization until up to 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (842):
- United States (269):
  - UAB St Vincents, Birmingham, Alabama
  - Eastern Shore Research Institute, Fairhope, Alabama
  - G and L Research LLC, Foley, Alabama
  - Alaska Heart and Vascular, Anchorage, Alaska
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Elite Clinical Studies, Phoenix, Arizona
  - HonorHealth Heart Group Deer Valley, Scottsdale, Arizona
  - Clinical Research Inst of Arizona, Sun City West, Arizona
  - Pima Heart And Vascular Clin Rch, Tucson, Arizona
  - ARcare Center for Clinical Research, Little Rock, Arkansas
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Central Cardiology Medical Center, Bakersfield, California
  - Alliance Clinical, Canoga Park, California
  - Inland Psychiatric Medical Group, Chino, California
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Triallogix, Fullerton, California
  - Diabetes Lipid Management Center, Huntington Beach, California
  - University of Calif Irvine Med Cntr, Irvine, California
  - UC San Diego Health, La Jolla, California
  - American Institute of Research, Los Angeles, California
  - Keck Medical Center USC, Los Angeles, California
  - University of California LA, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - San Diego Veterans Medical Center, San Diego, California
  - West Coast Research LLC, San Ramon, California
  - Helping Hands Medical Associates INC, Santa Ana, California
  - Syrentis Clinical Research, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - Stanford University Medical Center, Stanford, California
  - Manshadi Heart Institute, Stockton, California
  - Harbor UCLA Medical Center, Torrance, California
  - Blue Coast Research Center LLC, Vista, California
  - Interv Cardiology Med Grp, West Hills, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Rocky Mountain Regional VA Med Ctr, Aurora, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - d-b-a Greenwich Cardio Assoc, Greenwich, Connecticut
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Emerson Clinical Research Institute, Washington D.C., District of Columbia
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - Cardiovascular and Vein Center of Florida, Bradenton, Florida
  - Nova Clinical Research LLC, Bradenton, Florida
  - Bay Care Medical Group, Clearwater, Florida
  - Cardiology Research Associates, Daytona Beach, Florida
  - Hillcrest Medical Research, DeLand, Florida
  - Indago Research and Health Ctr Inc, Hialeah, Florida
  - National Research Institute, Hialeah, Florida
  - Sister Life Research Inc, Hialeah, Florida
  - Zenith Clinical Research, Hollywood, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - UF Health Science Center, Jacksonville, Florida
  - Baptist Heart Specialists, Jacksonville Beach, Florida
  - United Vein and Vascular Centers, Lake Worth, Florida
  - Infinite Clinical Research, Miami, Florida
  - A&A Research Group Inc, Miami, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - RM Medical Research Inc, Miami Lakes, Florida
  - FXM Clin Res Miramar LLC, Miramar, Florida
  - Advanced Research for Health Improvement LLC, Naples, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - CTMD Research, Palm Springs, Florida
  - Broward Research Center, Pembroke Pines, Florida
  - SEC Clinical Research, Pensacola, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Advanced Medical Research Center, St. Petersburg, Florida
  - New Tampa Health, Tampa, Florida
  - James A Haley Veterans Hospital, Tampa, Florida
  - BayCare Medical Group Inc, Tampa, Florida
  - Genesis Clinical Research, Tampa, Florida
  - BayCare Health System, Tampa, Florida
  - Ravessa Clinical Research, Tampa, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Javara Research, Fayetteville, Georgia
  - Northeast Georgia Medical Center, Gainsville, Georgia
  - Alta Pharmaceutical Research Center, Peachtree Corners, Georgia
  - Atlanta Heart Specialists LLC, Tucker, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Saltzer Health, Nampa, Idaho
  - Biofortis Research, Addison, Illinois
  - Endeavor Health Clinical Op- NCH, Arlington Heights, Illinois
  - Cedar Crosse Research Ct, Chicago, Illinois
  - Chicago Clinical Research Inst, Chicago, Illinois
  - Gateway Cardiology PC, Jerseyville, Illinois
  - Methodist Med Center Of Illinois, Peoria, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - Prairie Heart Institute, Springfield, Illinois
  - Elkhart Cardiology Group, Elkhart, Indiana
  - Franciscan Health Services Research Center, Indianapolis, Indiana
  - Witham Heart Partners, Lebanon, Indiana
  - The Heart Center of Lake County, Merrillville, Indiana
  - Cardiovascular Research Of Northwest Indiana, Llc, Munster, Indiana
  - Covenant Medical Center, Waterloo, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Midwest Heart and Vascular Spec, Overland Park, Kansas
  - Cotton O Neil Clinical Res Center, Topeka, Kansas
  - Ascension Via Christi Research, Wichita, Kansas
  - University of Kentucky College of Health Sciences, Lexington, Kentucky
  - U of Louisville Rudd Heart and Lung, Louisville, Kentucky
  - Christus Health Central Louisiana, Alexandria, Louisiana
  - Louisiana Cardiology Associates, Baton Rouge, Louisiana
  - Grace Research LLC, Bossier City, Louisiana
  - Cardiovascular Associates Research, Covington, Louisiana
  - Louisiana Heart Center Research, Covington, Louisiana
  - Avant Research Associates LLC, Crowley, Louisiana
  - Horizon Research Group of Opelousas LLC, Eunice, Louisiana
  - Cardiovascular Institute South ASC, Gray, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - CV Ins of the South, Lafayette, Louisiana
  - North Shore Heart and Vascular, Mandeville, Louisiana
  - Clinical Trials Management LLC, Mandeville, Louisiana
  - Omega Clinical Research, Metairie, Louisiana
  - Clinical Trials of America LA LLC, Monroe, Louisiana
  - Barnum Medical Research Inc, Natchitoches, Louisiana
  - Crescent City Physicians Inc, New Orleans, Louisiana
  - CV Ins of the South, Opelousas, Louisiana
  - Grace Research Llc, Shreveport, Louisiana
  - Louisiana Heart Center Research, Slidell, Louisiana
  - Southern Clinical Research, Zachary, Louisiana
  - Sinai Ct for Throm Res and Drug Dev, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants Llc, Beltsville, Maryland
  - Johns Hopkins University, Columbia, Maryland
  - Anderson Medical Research, Ft. Washington, Maryland
  - Javara Inc, Glenn Dale, Maryland
  - Capitol Cardiology Associates, Lanham, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Adventist HealthCare Shady Grove Medical Center, Rockville, Maryland
  - Tidal Health Peninsula Regional Inc, Salisbury, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - VA Boston Healthcare System, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - AA Medical Research Center, Flint, Michigan
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - McLaren Greater Lansing, Lansing, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Central Michigan University, Saginaw, Michigan
  - Providence Hospital Patient Care Research, Southfield, Michigan
  - Traverse Heart and Vascular, Traverse City, Michigan
  - Trinity Health Michigan Heart, Ypsilanti, Michigan
  - St Marys Medical Center, Duluth, Minnesota
  - University Of Minnesota, Minneapolis, Minnesota
  - North Memorial Heart and Vascular Institute, Robbinsdale, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Belzoni Clinical Research, Belzoni, Mississippi
  - Jackson Heart Clinic, Jackson, Mississippi
  - VAMC Research-G V Sonny Montgomery Clinic, Jackson, Mississippi
  - Cardiology Associates of North MS, Tupelo, Mississippi
  - Yazoo Clinical Research ., Yazoo City, Mississippi
  - Yazoo Clinical Research, Yazoo City, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Hospital, Springfield, Missouri
  - St Louis V A Medical Center, St Louis, Missouri
  - Gateway Cardiovascular Rsch Ctr Inc, St Louis, Missouri
  - Mercy South, St Louis, Missouri
  - St Louis Heart and Vascular, St Louis, Missouri
  - Physician Research Collaboration, Lincoln, Nebraska
  - VA Med NWI Endocrine Studies R151, Omaha, Nebraska
  - CCT Research, Omaha, Nebraska
  - Las Vegas Endocrinology, Henderson, Nevada
  - AB Clinical Trials, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Catholic Medical Center, Manchester, New Hampshire
  - Cooper University Health Care, Haddon Heights, New Jersey
  - New Jersey Heart, Linden, New Jersey
  - Garden State Heart Care, Manalapan, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Meridian Clinical Research, Binghamton, New York
  - Bassett Medical Center, Cooperstown, New York
  - Meridian Clinical Research LLC, Endwell, New York
  - NYU Langone Hlth Card Assoc, Mineola, New York
  - Weill Cornell Medical Center, New York, New York
  - Icahn School of Med at Mt Sinai, New York, New York
  - Northport VA Medical Center, Northport, New York
  - Rochester Clinical Research, Rochester, New York
  - State Uni of NY at Stony Brook, Stony Brook, New York
  - Westchester Medical Center, Valhalla, New York
  - Novant Health Heart Vas Inst, Charlotte, North Carolina
  - Tryon Medical Partners PLLC, Charlotte, North Carolina
  - Lucas Research, Morehead City, North Carolina
  - NC Heart and Vascular Research LLC, Raleigh, North Carolina
  - Accellacare of Salisbury, Salisbury, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Altru Health Research Dept., Grand Forks, North Dakota
  - Akron Hospital Summa Health System, Akron, Ohio
  - Velocity Clin Research Springdale, Cincinnati, Ohio
  - University Of Cincinnati, Cincinnati, Ohio
  - Univ Hosp Cleveland Medical Center, Cleveland, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Rama Research LLC, Marion, Ohio
  - Heart House Research Foundation, Springfield, Ohio
  - Mercy Health St Vincent Med Ctr, Toledo, Ohio
  - Premier Cardiovascular Institute, Vandalia, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Samaritan Cardiology, Corvallis, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Independence Health System Cardiovascular Consultants, Butler, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Frontier Clinical Research LLC, Smithfield, Pennsylvania
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - Medical Univ Of South Carolina, Charleston, South Carolina
  - Columbia Heart Clinic, Columbia, South Carolina
  - Columbia VA Health Care System, Columbia, South Carolina
  - Bon Secours Medical Group, Greenville, South Carolina
  - Prisma Health Upstate, Greenville, South Carolina
  - Trident Cardiology, Ladson, South Carolina
  - Family Medicine of Sayebrook, Myrtle Beach, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - North Central Heart, Sioux Falls, South Dakota
  - Wellmont CVA Heart Institute, Greenville, Tennessee
  - Apex Cardiology Research Associates of Jackson, Jackson, Tennessee
  - The Jackson Clinic PA, Jackson, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Accellacare, Knoxville, Tennessee
  - Memphis Cardiology and Vein Ct, Memphis, Tennessee
  - Cardiovascular Res of Knoxville LLC, Powell, Tennessee
  - Tennessee Center For Clinical Trials, Tullahoma, Tennessee
  - PharmaTex Research LLC, Amarillo, Texas
  - North Hills Medical Research Inc, Bedford, Texas
  - Javara Research, Conroe, Texas
  - VA North Texas Health Care System, Dallas, Texas
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Research Institute of Dallas PA, Dallas, Texas
  - Texas Health Physicians Group, Dallas, Texas
  - SW Family Medicine Associates, Dallas, Texas
  - Alina clinical trials, Dallas, Texas
  - David Turbay MD PLLC, El Paso, Texas
  - Texas Health Physicians Group, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - UT Physicians Memorial Hermann, Houston, Texas
  - Orion Medical, Houston, Texas
  - Village Medical Village MD S Tx, Houston, Texas
  - FMC Science, Lampasas, Texas
  - East Texas Research Associates Inc., Livingston, Texas
  - CardioVoyage LLC, McKinney, Texas
  - Discovery Clinical Trials, Pflugerville, Texas
  - Heartplace-Plano, Plano, Texas
  - University of Texas Health Science Ctr, San Antonio, Texas
  - South Texas Cardiovascular Consultants PLLC, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Javara Research, Stephenville, Texas
  - Privia Medical Group Gulf Coast, Sugarland, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Burke Internal Medicine and Research, Burke, Virginia
  - Javara Research, Forest, Virginia
  - Heart Care Associates P C, Hopewell, Virginia
  - York Clinical Research, Norfolk, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Virginia Mason Medical Centre, Seattle, Washington
  - Swedish Medical Center-Cardiovascular Research, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Universal Research Group LLC, Tacoma, Washington
  - Confluence Health Hospital, Wenatchee, Washington
- Argentina (20):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, San Martín, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Formosa, Formosa Province
  - Novartis Investigative Site, Posadas, Misiones Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, San Miguel Tucuman, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Santa Fe
- Australia (16):
  - Novartis Investigative Site, Botany, New South Wales
  - Novartis Investigative Site, New Lambton Heights, New South Wales
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, Milton, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Leabrook, South Australia
  - Novartis Investigative Site, Woodville South, South Australia
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Geelong, Victoria
  - Novartis Investigative Site, Malvern East, Victoria
  - Novartis Investigative Site, Richmond, Victoria
  - Novartis Investigative Site, Joondalup, Western Australia
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Liverpool
- Austria (2):
  - Novartis Investigative Site, Braunau am Inn
  - Novartis Investigative Site, Graz
- Belgium (13):
  - Novartis Investigative Site, Genk, Limburg
  - Novartis Investigative Site, Yvoir, Namur
  - Novartis Investigative Site, Kortrijk, West-Vlaanderen
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, La Louvière
  - Novartis Investigative Site, Ronse
- Brazil (20):
  - Novartis Investigative Site, Maceió, Alagoas
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Canoas, Rio Grande do Sul
  - Novartis Investigative Site, Pelotas, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Aracaju, Sergipe
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, Sao Jose Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Campinas
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, São Paulo
- Bulgaria (18):
  - Novartis Investigative Site, Sandanski, Blagoevgrad
  - Novartis Investigative Site, Rousse, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Stara Zagora, Bulgaria
  - Novartis Investigative Site, Burgas, Burgas
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Haskovo
  - Novartis Investigative Site, Kyustendil
  - Novartis Investigative Site, Montana
  - Novartis Investigative Site, Pernik
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sliven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stamboliyski
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Veliko Tarnovo
- Canada (24):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, North Vancouver, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Sydney, Nova Scotia
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Guelph, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Oakville, Ontario
  - Novartis Investigative Site, Peterborough, Ontario
  - Novartis Investigative Site, Sarnia, Ontario
  - Novartis Investigative Site, Scarborough Village, Ontario
  - Novartis Investigative Site, Stoufville, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saint-Jérôme, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Terrebonne, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Chile (7):
  - Novartis Investigative Site, La Serena, Coquimbo Region
  - Novartis Investigative Site, Osorno, Los Lagos Region
  - Novartis Investigative Site, Temuco, Región de la Araucanía
  - Novartis Investigative Site, Victoria, Región de la Araucanía
  - Novartis Investigative Site, Viña del Mar, Región de Valparaíso
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
  - Novartis Investigative Site, Santiago
- China (35):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Foshan, Guangdong
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Jingzhou, Hubei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Hohhot, Inner Mongolia
  - Novartis Investigative Site, Changzhou, Jiangsu
  - Novartis Investigative Site, Jiangyin, Jiangsu
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Xuzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Pingxiang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Lishui, Zhejiang
  - Novartis Investigative Site, Taizhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Xiamen
- Colombia (10):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Manizales, Caldas Department
  - Novartis Investigative Site, Barranquilla, Colombia
  - Novartis Investigative Site, Cali, Colombia
  - Novartis Investigative Site, Cartagena, Departamento de Bolívar
  - Novartis Investigative Site, Pereira, Risaralda Department
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Floridablanca
- Croatia (9):
  - Novartis Investigative Site, Krapinske Toplice, Croatia
  - Novartis Investigative Site, Slavonski Brod, Croatia
  - Novartis Investigative Site, Zagreb, Croatia
  - Novartis Investigative Site, Čakovec
  - Novartis Investigative Site, Opatija
  - Novartis Investigative Site, Osijek
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Split
  - Novartis Investigative Site, Zagreb
- Czechia (20):
  - Novartis Investigative Site, Louny, Czech Republic
  - Novartis Investigative Site, Bedihošť
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Český Krumlov
  - Novartis Investigative Site, Hodonín
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Mariánské Lázně
  - Novartis Investigative Site, Náchod
  - Novartis Investigative Site, Ostrava
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Polička
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Přerov
  - Novartis Investigative Site, Příbram
  - Novartis Investigative Site, Slaný
  - Novartis Investigative Site, Svitavy
  - Novartis Investigative Site, Třebíč
  - Novartis Investigative Site, Uherské Hradiště
  - Novartis Investigative Site, Zlín
- Denmark (9):
  - Novartis Investigative Site, Herning, Central Jutland
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Glostrup Municipality
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Hjørring
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Svendborg
  - Novartis Investigative Site, Viborg
- Estonia (3):
  - Novartis Investigative Site, Pärnu
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (4):
  - Novartis Investigative Site, Kuopio, Northern Savonia
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Jyväskylä
  - Novartis Investigative Site, Turku
- France (29):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Béziers
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Cholet
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Le Coudray
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Orléans
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pau
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tourcoing
  - Novartis Investigative Site, Valenciennes
  - Novartis Investigative Site, Villeneuve-d'Ascq
- Greece (4):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Larissa
  - Novartis Investigative Site, Thessaloniki
- Hungary (19):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Oroshaza, Csongrád megye
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest, Pest County
  - Novartis Investigative Site, Baja
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Balatonfüred
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kalocsa
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Komárom
  - Novartis Investigative Site, Nagykanizsa
  - Novartis Investigative Site, Orosháza
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szekszárd
  - Novartis Investigative Site, Szolnok
  - Novartis Investigative Site, Zalaegerszeg
- Iceland (2):
  - Novartis Investigative Site, Kopavogur
  - Novartis Investigative Site, Reykjavik
- India (32):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Guntur, Andhrapradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Belagavi, Karnataka
  - Novartis Investigative Site, Manipal, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Kozhikode, Kerala
  - Novartis Investigative Site, Indore, Madhyapradesh
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Secunderabad, Telangana
  - Novartis Investigative Site, Aligarh, Uttar Pradesh
  - Novartis Investigative Site, Ghaziabad, Uttar Pradesh
  - Novartis Investigative Site, Kanpur, Uttar Pradesh
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
  - Novartis Investigative Site, Dehradun, Uttarakhand
  - Novartis Investigative Site, Dehradun, Uttrakhand
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, New Delhi
  - Novartis Investigative Site, Puducherry
  - Novartis Investigative Site, Uttarakhand
- Israel (8):
  - Novartis Investigative Site, Ashdod
  - Novartis Investigative Site, Holon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Nahariya
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Sefad
  - Novartis Investigative Site, Ẕerifin
- Italy (13):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Grosseto, GR
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Torino, TO
- Japan (12):
  - Novartis Investigative Site, Toyota, Aichi-ken
  - Novartis Investigative Site, Chikushino-shi, Fukuka
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Komatsu, Ishikawa-ken
  - Novartis Investigative Site, Fujisawa, Kanagawa
  - Novartis Investigative Site, Odawara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Nagaoka, Niigata
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Kawaguchi, Saitama
- Novartis Investigative Site, Nairobi, Kenya
- Latvia (6):
  - Novartis Investigative Site, Liepāja, LV
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Kuldīga
  - Novartis Investigative Site, Riga
  - Novartis Investigative Site, Valmiera
- Lithuania (7):
  - Novartis Investigative Site, Kaunas, Kaunas County
  - Novartis Investigative Site, Klaipėda, Klaipėda County
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Šiauliai, LTU
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Panevezys
  - Novartis Investigative Site, Vilnius
- Malaysia (5):
  - Novartis Investigative Site, Alor Star, Kedah
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, Kuala Lumpur, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Mauritius (2):
  - Novartis Investigative Site, Solferino Phoenix, Mauritius
  - Novartis Investigative Site, Phoenix
- Mexico (12):
  - Novartis Investigative Site, Aguascalientes, Aguascalientes
  - Novartis Investigative Site, Tlalnepantla, Edo de Mexico
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, Acapulco
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Chihuahua City
  - Novartis Investigative Site, Durango
  - Novartis Investigative Site, Guadalajara
  - Novartis Investigative Site, Xalapa
- Netherlands (20):
  - Novartis Investigative Site, Meppel, Drenthe
  - Novartis Investigative Site, Doetinchem, Gelderland
  - Novartis Investigative Site, Nijmegen, Gelderland
  - Novartis Investigative Site, Tiel, Gelderland
  - Novartis Investigative Site, Nijmegen, Gerlderland
  - Novartis Investigative Site, Breda, North Brabant
  - Novartis Investigative Site, Tilburg, North Brabant
  - Novartis Investigative Site, Alkmaar, North Holland
  - Novartis Investigative Site, Amstelveen, North Holland
  - Novartis Investigative Site, Amsterdam, North Holland
  - Novartis Investigative Site, Heemstede, North Holland
  - Novartis Investigative Site, Deventer, Overijssel
  - Novartis Investigative Site, Leeuwarden, Provincie Friesland
  - Novartis Investigative Site, Sneek, Provincie Friesland
  - Novartis Investigative Site, Groningen, Provincie Groningen
  - Novartis Investigative Site, Leiden, South Holland
  - Novartis Investigative Site, Leiderdorp, South Holland
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Gouda
  - Novartis Investigative Site, Venlo
- New Zealand (7):
  - Novartis Investigative Site, Grafton, Auckland
  - Novartis Investigative Site, Christchurch, Christchurch
  - Novartis Investigative Site, Dunedin, NZW
  - Novartis Investigative Site, Auckland
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Lower Hutt
- Norway (7):
  - Novartis Investigative Site, Nordbyhagen, Oslo County
  - Novartis Investigative Site, Stavanger, Stavanger
  - Novartis Investigative Site, Arendal
  - Novartis Investigative Site, Drammen
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Skedsmokorset
  - Novartis Investigative Site, Tromsø
- Philippines (4):
  - Novartis Investigative Site, Iloilo City, Iloilo
  - Novartis Investigative Site, San Fernando City, Pampanga
  - Novartis Investigative Site, Quezon
  - Novartis Investigative Site, San Juan City
- Poland (20):
  - Novartis Investigative Site, Nowy Targ, Lesser Poland Voivodeship
  - Novartis Investigative Site, Ostrołęka, Masovian Voivodeship
  - Novartis Investigative Site, Sosnowiec, Silesian Voivodeship
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Kłodzko
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Ostrowiec Swietok
  - Novartis Investigative Site, Puławy
  - Novartis Investigative Site, Ruda Śląska
  - Novartis Investigative Site, Skierniewice
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Włocławek
  - Novartis Investigative Site, Zamość
- Portugal (11):
  - Novartis Investigative Site, Alcabideche
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Carnaxide
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Guimarães
  - Novartis Investigative Site, Leiria
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Santa Maria da Feira
  - Novartis Investigative Site, Vila Nova de Gaia
  - Novartis Investigative Site, Vila Real
- Puerto Rico (5):
  - Advanced Clinical Research LLC, Bayamón
  - Research and Cardiovascular Corp, Ponce
  - Latin Clinical Trial Center Inc, San Juan
  - Advance Medical Research Center, San Juan
  - Barbara Diaz Hernandez Research Inc, San Juan
- Romania (13):
  - Novartis Investigative Site, Piteşti, Argeş
  - Novartis Investigative Site, Oradea, Jud Bihor
  - Novartis Investigative Site, Baia Mare, Maramureş
  - Novartis Investigative Site, Târgu Mureş, Mureș County
  - Novartis Investigative Site, Brăila, ROM
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Caracal
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Iași
  - Novartis Investigative Site, Târgu Mureş
  - Novartis Investigative Site, Timișoara
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- Serbia (11):
  - Novartis Investigative Site, Belgrade, Serbia
  - Novartis Investigative Site, Kamenitz, Serbia
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Ćuprija
  - Novartis Investigative Site, Kragujevac
  - Novartis Investigative Site, Leskovac
  - Novartis Investigative Site, Niš
  - Novartis Investigative Site, Smederevo
  - Novartis Investigative Site, Subotica
  - Novartis Investigative Site, Vranje
  - Novartis Investigative Site, Zaječar
- Singapore (2):
  - Novartis Investigative Site, Singapore, Singapore
  - Novartis Investigative Site, Singapore
- Slovakia (15):
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Moldava nad Bodvou
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Piešťany
  - Novartis Investigative Site, Považská Bystrica
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Rožňava
  - Novartis Investigative Site, Žilina
- Slovenia (4):
  - Novartis Investigative Site, Celje
  - Novartis Investigative Site, Ljubljana
  - Novartis Investigative Site, Ptuj
  - Novartis Investigative Site, Slovenj Gradec
- South Africa (15):
  - Novartis Investigative Site, Raslouw, Centurion
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Germiston, Gauteng
  - Novartis Investigative Site, Pretoria, Gauteng
  - Novartis Investigative Site, Soweto, Gauteng
  - Novartis Investigative Site, Vereeniging, Gauteng
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, George, Western Cape
  - Novartis Investigative Site, Paarl, Western Cape
  - Novartis Investigative Site, Cape Town, ZAF
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Midrand
  - Novartis Investigative Site, Pretoria
  - Novartis Investigative Site, Worcester
- South Korea (14):
  - Novartis Investigative Site, Daegu, Dalseo gu
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Jinju, Gyeongsangnam-do
  - Novartis Investigative Site, Yangsan, Gyeongsangnam-do
  - Novartis Investigative Site, Incheon, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Spain (34):
  - Novartis Investigative Site, Ferrol, A Coruna
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Mallorca, Balearic Islands
  - Novartis Investigative Site, Palma, Balearic Islands
  - Novartis Investigative Site, el Prat de Llobregat, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Sant Joan Despí, Barcelona
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, Jerez de la Frontera, Cadiz
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, San Sebastian Reyes, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Utrera, Sevilla
  - Novartis Investigative Site, Reus, Tarragona
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Almería
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, Huelva
  - Novartis Investigative Site, Las Palmas GC
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Valladolid
  - Novartis Investigative Site, Zaragoza
- Sweden (8):
  - Novartis Investigative Site, Stockholm, SE
  - Novartis Investigative Site, Gothenburg, Västra Götaland County
  - Novartis Investigative Site, Falun
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Västerås
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Thailand (5):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Muang, Thailand
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Muang
- Turkey (Türkiye) (9):
  - Novartis Investigative Site, Izmir, Balcova
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Istanbul, Kartal
  - Novartis Investigative Site, Bursa, Nilufer
  - Novartis Investigative Site, Konya, Selcuklu
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Adana, Yuregir
  - Novartis Investigative Site, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com